CLINICAL TRIAL: NCT00796367
Title: A Phase 3, Double-Blind, Placebo-Controlled, Multicenter Extension Study (From Study OB-303 [NCT00553787]) to Determine the Safety and Efficacy Of VI-0521 for the Long-Term Treatment Of Obesity in Adults With Obesity-Related Co-Morbid Conditions.
Brief Title: A Safety and Efficacy Study of VI-0521 to Evaluate the Long Term Treatment of Obesity in Adults With Obesity-Related Co-Morbid Conditions. An Extension Study of Protocol OB-303 (NCT00553787)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OB-305
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Qsymia; Qnexa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- VI-0521 Mid (Experimental): 7.5 mg phentermine and 46 mg topiramate
  Interventions: Drug: VI-0521
- VI-0521 Top (Experimental): 15 mg phentermine and 92 mg topiramate
  Interventions: Drug: VI-0521

INTERVENTIONS:
Drug: VI-0521 — 7.5 mg phentermine and 46 mg topiramate
  Other Names: Qsymia; Qnexa; PHEN/TPM
  Arms: VI-0521 Mid
Drug: Placebo — placebo
  Arms: Placebo
Drug: VI-0521 — 15 mg phentermine and 92 mg topiramate
  Other Names: Qsymia; Qnexa; PHEN/TPM
  Arms: VI-0521 Top

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of VI-0521 compared to placebo for the treatment of overweight and obesity in adults who have completed study OB-303 (NCT00553787) at selected study sites. This is an extension study of protocol OB-303 (NCT00553787).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment into this study, subjects must meet all of the following criteria:

* Completion of study OB-303 (NCT00553787) on treatment and compliance with all protocol requirements
* Written informed consent
* Female subjects of childbearing potential must be using adequate contraception, defined as double-barrier methods, stable hormonal contraception plus single barrier method, or tubal ligation. Female subjects are considered to be of childbearing potential unless they have undergone a hysterectomy or bilateral oophorectomy, are ≥55 years of age and experienced spontaneous cessation of menses for at least 1 year, or have a documented follicle-stimulating hormone level ≥40 IU/L
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects will not be included in the study if they meet any of the following:

* Body mass index ≤22 kg/m2 at the completion of study OB-303
* Off study medication at completion of study OB-303 (NCT00553787) for longer than 4 weeks continuously due to an event-driven holiday, or off study medication with no plans to restart
* Development of any condition during study OB-303 (NCT00553787) that, in the opinion of the investigator, would contraindicate the administration of study medication, affect compliance, interfere with study evaluations, or confound the interpretation of study results
* Participation in a formal weight loss program (including: Weight Watchers and related dietary/lifestyle intervention programs; prepared food programs; prescribed or over the counter weight loss medications; dietary supplement or herbal preparations, teas, or tinctures intended for weight loss; or any supervised fast or very low calorie diet).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, Study Director — VIVUS LLC

REFERENCES:
- [Derived] Guo F, Garvey WT. Cardiometabolic Disease Staging Predicts Effectiveness of Weight-Loss Therapy to Prevent Type 2 Diabetes: Pooled Results From Phase III Clinical Trials Assessing Phentermine/Topiramate Extended Release. Diabetes Care. 2017 Jul;40(7):856-862. doi: 10.2337/dc17-0088. Epub 2017 Apr 28. PMID 28455281
- [Derived] Garvey WT, Ryan DH, Look M, Gadde KM, Allison DB, Peterson CA, Schwiers M, Day WW, Bowden CH. Two-year sustained weight loss and metabolic benefits with controlled-release phentermine/topiramate in obese and overweight adults (SEQUEL): a randomized, placebo-controlled, phase 3 extension study. Am J Clin Nutr. 2012 Feb;95(2):297-308. doi: 10.3945/ajcn.111.024927. Epub 2011 Dec 7. PMID 22158731
- See also: VIVUS company website — http://www.vivus.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were from OB-303 (NCT00553787)
Groups:
- VI-0521 Mid: VI-0521 7.5 mg PHEN/46 mg TPM
- VI-0521 Top: VI-0521 15 mg PHEN/92 mg TPM
Period: Overall Study
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Started | 227 | 154 (one participant signed ICF but withdrew from study prior to first dosing in OB-305) | 295
Completed | 197 | 129 | 248
Not Completed | 30 | 25 | 47
Not completed — Adverse Event | 6 | 4 | 7
Not completed — Lost to Follow-up | 5 | 4 | 21
Not completed — Withdrawal by Subject | 9 | 11 | 12
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — non compliance | 3 | 1 | 1
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Requirement for restricted medication | 2 | 0 | 2
Not completed — other | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top | Total
Number analyzed (Participants) | 227 | 153 | 295 | 675
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.8) | 52.2 (10.6) | 51.2 (10.4) | 51.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 106 | 195 | 448
  Male | 80 | 47 | 100 | 227
Region of Enrollment [Number; unit: participants]
  United States | 227 | 153 | 295 | 675

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change at End of Treatment, Week 108.
Time Frame: From baseline to end of treatment
Population: Intent-to-Treat Last observation carried forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent weight loss
Groups:
- VI-0521 Mid: VI-0521 7.5 mg phentermine/46 mg topiramate
- VI-0521 Top: VI-0521 15 mg phentermine/92 mg topiramate
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Number analyzed (Participants) | 227 | 153 | 295
percent weight loss | -1.8 (0.55) | -9.32 (0.67) | -10.5 (0.5)
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Top; No formal calculation of sample size was conducted due to being an extension study of OB-303 (NCT00553787); Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 8.71, 95% CI 2-sided [7.39 to 10.03], Standard Error of Mean 0.673
Statistical Analysis 2: Comparison: Placebo vs VI-0521 Mid; No formal calculation of sample size was conducted due to being an extension study of OB-303 (NCT00553787); Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 7.52, 95% CI 2-sided [5.95 to 9.09], Standard Error of Mean 0.799
Statistical Analysis 3: Comparison: VI-0521 Mid vs VI-0521 Top; No formal calculation of sample size was conducted due to being an extension study of OB-303 (NCT00553787); Test type: Superiority or Other; p = 0.1189, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-0.31 to 2.68], Standard Error of Mean 0.760

2. Primary Outcome: Percentage of Subjects With at Least 5% Weight Loss at End of Treatment, Week 108.
Time Frame: Baseline to End of Treatment
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Number; unit: percent participants
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Number analyzed (Participants) | 227 | 153 | 295
percent participants | 30 | 75.2 | 79.3
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Top; No formal calculation of sample size was conducted due to being an extension study of OB-303 (NCT00553787); Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 9.4, 95% CI 2-sided [6.24 to 14.16], Standard Error of Mean 1.97
Statistical Analysis 2: Comparison: Placebo vs VI-0521 Mid; No formal calculation of sample size was conducted due to being an extension study of OB-303 (NCT00553787); Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 6.99, 95% CI 2-sided [4.36 to 11.19], Standard Error of Mean 1.68
Statistical Analysis 3: Comparison: VI-0521 Mid vs VI-0521 Top; No formal calculation of sample size was conducted due to being an extension study of OB-303 (NCT00553787); Test type: Superiority or Other; p = 0.2169, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.84 to 2.15], Standard Error of Mean 0.32

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Serious Adverse Events (participants affected / at risk) | 9/227 | 4/153 | 13/295
Other Adverse Events (participants affected / at risk) | 182/227 | 111/153 | 234/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=227) | VI-0521 Mid (N=153) | VI-0521 Top (N=295)
ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
hemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
transient ischemic attack (Nervous system disorders) | 0 | 1 | 0
cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
ischemic stroke (Nervous system disorders) | 0 | 0 | 1
depression (Psychiatric disorders) | 1 | 0 | 0
peptic ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
nephritic syndrome (Renal and urinary disorders) | 1 | 0 | 0
renal failure, acute (Renal and urinary disorders) | 0 | 0 | 2
pneumonia (Infections and infestations) | 1 | 0 | 1
appendicitis (Infections and infestations) | 1 | 0 | 2
pyelonephritis (Infections and infestations) | 0 | 1 | 0
influenza (Infections and infestations) | 0 | 0 | 1
mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
hypotension (Vascular disorders) | 1 | 0 | 0
drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
serositis (General disorders) | 1 | 0 | 0
myocardial infarction (Cardiac disorders) | 0 | 1 | 0
acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
acute cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=227) | VI-0521 Mid (N=153) | VI-0521 Top (N=295)
upper respiratory tract infection (Infections and infestations) | 42 | 26 | 45
nasopharyngitis (Infections and infestations) | 26 | 13 | 26
sinusitis (Infections and infestations) | 18 | 12 | 28
urinary tract infection (Infections and infestations) | 13 | 14 | 18
influenza (Infections and infestations) | 8 | 10 | 19
bronchitis (Infections and infestations) | 7 | 8 | 10
constipation (Gastrointestinal disorders) | 7 | 11 | 12
nausea (Gastrointestinal disorders) | 4 | 10 | 4
arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 7 | 16
back pain (Musculoskeletal and connective tissue disorders) | 7 | 9 | 15
insomnia (Psychiatric disorders) | 8 | 9 | 11
procedural pain (Injury, poisoning and procedural complications) | 4 | 8 | 14
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 4 | 6
pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 3 | 5
Gastroenteritis (Infections and infestations) | 6 | 2 | 9
gastroenteritis viral (Infections and infestations) | 6 | 4 | 4
ear infection (Infections and infestations) | 2 | 3 | 7
tooth abscess (Infections and infestations) | 4 | 4 | 4
pneumonia (Infections and infestations) | 4 | 4 | 3
viral infection (Infections and infestations) | 3 | 2 | 6
tooth infection (Infections and infestations) | 1 | 3 | 4
oral herpes (Infections and infestations) | 2 | 3 | 2
osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 7
muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4 | 6
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6
diarrhea (Gastrointestinal disorders) | 3 | 3 | 11
tooth ache (Gastrointestinal disorders) | 5 | 4 | 2
abdominal pain (Gastrointestinal disorders) | 5 | 0 | 3
hemorrhoids (Gastrointestinal disorders) | 1 | 1 | 6
vomiting (Gastrointestinal disorders) | 2 | 4 | 1
abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 0
joint sprain (Injury, poisoning and procedural complications) | 4 | 5 | 7
muscle strain (Injury, poisoning and procedural complications) | 4 | 6 | 6
contusion (Injury, poisoning and procedural complications) | 2 | 3 | 7
cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 10
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 8
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3
headache (Nervous system disorders) | 6 | 4 | 12
paresthesia (Nervous system disorders) | 0 | 1 | 10
depression (Psychiatric disorders) | 2 | 3 | 10
anxiety (Psychiatric disorders) | 3 | 3 | 6
diabetes mellitus (Metabolism and nutrition disorders) | 7 | 1 | 3
dyslipidemia (Metabolism and nutrition disorders) | 6 | 2 | 0
weight increased (Investigations) | 5 | 0 | 7
hemoglobin decreased (Investigations) | 2 | 3 | 0
abdominal bruit (Investigations) | 0 | 3 | 1
edema peripheral (General disorders) | 7 | 0 | 12
eye pain (Eye disorders) | 2 | 4 | 4
hypertension (Vascular disorders) | 9 | 2 | 10
seasonal allergy (Immune system disorders) | 2 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.